CLINICAL TRIAL: NCT04633798
Title: Evaluation of the Efficacy of Intense Pulse Light Combined With Lipiflow in the Treatment of Meibomian Gland Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aier School of Ophthalmology, Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHAIER2020IRB04
Record Dates: First submitted 2020-05-20; First posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPL/Lipiflow (Experimental): the group in which patients treated with IPL combined with lipiflow
  Interventions: Procedure: IPL/Lipiflow
- IPL/MGX (Active Comparator): the group in which patients treated with IPL combined with meibomian gland massage
  Interventions: Procedure: IPL/MGX

INTERVENTIONS:
Procedure: IPL/Lipiflow — To treat patients with MGD using intense pulsed light combined with lipiflow
  Arms: IPL/Lipiflow
Procedure: IPL/MGX — To treat patients with MGD using intense pulsed light combined with meibomian gland massage
  Arms: IPL/MGX

SUMMARY:
To compare the effect of IPL combined with lipiflow and IPL combined with meibomian gland massage in treating meibomian gland dysfunction of different degrees ,focusing on effective rate, lasting time and changes of meibomian gland function and morphology.

DETAILED DESCRIPTION:
To divide all participants into two groups, group one treated with IPL combined with Lipiflow and group two treated with IPL combined with meibomian gland massage.The following parameters were recorded after treatment: the effective rate, lasting time and changes of meibomian gland function and morphology.All parameters were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* patients with meibomian gland dysfunction
* patients with ocular discomfort
* skin type:FitzpatricⅠ-Ⅳ

Exclusion Criteria:

* patients with acute ocular inflammation
* eye surgery history in the last 12 months
* patients who have received IPL or Lipiflow in the last 12 months
* patients who wear contact lens in last one month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2020-12-21 (Estimated); Study Completion 2020-12-21 (Estimated)

PRIMARY OUTCOMES:
ocular surface disease index(OSDI) | 6 months
  The OSDI is assessed on a scale of 0 to 100,with higher scores representing greater disability
meibomian gland expressibility score and meibum quality score | 6 months
  The score is on a scale of 0 to 6.The higher scores, the severity of the meibomian gland function(the highest score is 6 and the lowest score is 0)
meibomian gland dropout score | 6 months
  the higher scores, the severity of the meibomian gland morphology(The highest score is 6 and the lowest score is 0)
Breakup time | 6 months
  the shorter time, the poorer of the tear film stability

CONTACTS AND LOCATIONS:
Overall Officials: Yan Chen, doctor, Principal Investigator — Shanghai aier eys hospital

IPD SHARING:
Plan to Share IPD: No